CLINICAL TRIAL: NCT01256788
Title: Prospective Randomized Study Evaluating Clinical Effectiveness of Post-op Treatment With Hyaluronic Acid Injections in Degenerative Joint Disease & Meniscal Tears
Brief Title: Post-op Treatment With Hyaluronic Acid Injections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insurance now covers post-op HA injections, drastically decreasing enrollment.
Sponsor: The Hawkins Foundation (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00007133
Record Dates: First submitted 2010-12-06; First posted 2010-12-09 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Meniscus Tear; Chondropathy/Degenerative Joint Disease (DJD)
Keywords: viscosupplementation; meniscus tear; degenerative joint disease
MeSH Terms: conditions — Cartilage Diseases; Joint Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The two treatment groups were:
  1. Received saline injection
  2. Received viscosupplementation injection
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viscosupplementation (Experimental): Hyaluronic acid injection
  Interventions: Device: Euflexxa
- Saline injection (Placebo Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Device: Euflexxa — 4 injections of 2ml of Euflexxa
  Arms: Viscosupplementation
Other: Saline — 4 injections of 3 ml of sterile saline
  Arms: Saline injection

SUMMARY:
This study will look at patients with post-operative treatment of a meniscal tear or degenerative joint disease (degenerative arthritis). They will be randomized into one of three groups: Euflexxa injection, saline (placebo) injection, or no injection. Those who are randomized into the injection group will receive a series of three injections (one a week for 3 weeks), then a "booster" injection at 6 months post-op. Several questionnaires will be given after the first set of injections, then again at a one year follow-up.

The hypothesis is that patients receiving hyaluronic acid injections will have better pain and function scores as compared with placebo and no further treatment at all time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients in post-op stage of treatment for meniscal tears or chondropathy/DJD
* Over 40 years of age
* A daily knee pain above 20mm on a 100mm visual analogue scale

Exclusion Criteria:

* Previous recipient of viscosupplementation injections
* Had rheumatoid arthritis or other inflammatory arthritis
* Had intra-articular steroid injections within the previous 2 months
* Invasive knee procedures within the past 6 months
* Contraindications to hyaluronate (an allergy)
* Medications that could interfere with the planned interventions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pace, MD, Study Chair — Greenville Hospital System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment: No injection - pain/function questionnaires only through 1 year
Period: Overall Study
Arm/Group | Viscosupplementation | Saline Injection | No Treatment
Started | 12 | 14 | 8
Completed | 7 | 6 | 5
Not Completed | 5 | 8 | 3
Not completed — Lost to Follow-up | 5 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- No Treatment: No injections given
- Total: Total of all reporting groups
Arm/Group | Viscosupplementation | Saline Injection | No Treatment | Total
Number analyzed (Participants) | 12 | 14 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 7 | 30
  >=65 years | 2 | 1 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (7.8) | 55.5 (8.7) | 56 (8.46) | 56 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 5 | 19
  Male | 4 | 8 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Tegner Activity Level Scale Score
Description: The Tegner Scoring system is a numeric scale range from 1 to 10, with each value indicating the ability to perform a specific activity. The scoring system is ordinal in nature and reflects lower to higher levels of activity participation, with higher numbers indicating a higher level of function.
Time Frame: 1 yr postop
Population: Study ended earlier due to problematic recruitment issues related to a change in insurance payments. Each treatment groups experienced lost to follow up, therefore the number of participants analyzed is smaller than the number of participants enrolled for each group.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- No Treatment: Patients did not receive neither viscosupplementation nor saline.
Arm/Group | Viscosupplementation | Saline Injection | No Treatment
Number analyzed (Participants) | 7 | 4 | 3
score on a scale | 2.5781 [1 to 5] | 3.5 [1 to 5] | 3 [1 to 5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Viscosupplementation | Saline Injection | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/8

LIMITATIONS AND CAVEATS:
Early termination due to new insurance coverage for post-operative knee viscosupplementation leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No